CLINICAL TRIAL: NCT03540589
Title: Distraction and Vibration for Minimizing Pain During Childhood Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Marcio Manozzo Boniatti, Professor, Hospital Nossa Senhora da Conceicao
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PCV-001
Record Dates: First submitted 2018-04-23; First posted 2018-05-30 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Pain Due to Childhood Vaccination
MeSH Terms: interventions — Osteogenesis, Distraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Video distraction (Experimental): A video will be available as soon as the child is randomized to this group, thus enabling the child to become more involved with distraction. A tablet will be delivered to the parents in the reception room to be viewed by the child before entering the vaccine room. After entering the room, the parents will keep the child entertained with the videos. There will be several videos, and it may be optional for the parents to choose according to their preferences.
  Interventions: Behavioral: Distraction
- Vibration device (Experimental): Buzzy® specific vibration device will be placed by the professional or caregiver at the application site, 15 to 45 seconds before the procedure.
  Interventions: Device: Buzzy specific vibration device
- Distraction plus vibration (Experimental): Combination of the two interventions described above
  Interventions: Device: Buzzy specific vibration device; Behavioral: Distraction
- Usual care (No Intervention): The vaccine will be carried out according to the routine of the Vaccine Center. Lidocaine plus prilocaine, non-nutritive sucking or breastfeeding may be used.

INTERVENTIONS:
Device: Buzzy specific vibration device — It is a device that produces vibration
  Arms: Distraction plus vibration; Vibration device
Behavioral: Distraction — The distraction will be obtained through tablet with videos
  Arms: Distraction plus vibration; Video distraction

SUMMARY:
Vaccine pain control is one of the actions suggested to support the delivery of vaccines that are on a vaccine schedule, since pain and anxiety associated with vaccines are among the main reasons why children and their parents fail to do them properly. Thus, it is very important to investigate which interventions can bring greater benefit in the control of pain.This is a randomized clinical trial aiming to assess the impact of video distraction and vibration device on pain during the vaccination of children between one and three years.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 year and 3 years, 11 months and 29 days of life.
* Be accompanied by legal guardian.
* Apply only one injectable vaccine at the time of the research.

Exclusion Criteria:

* Refuses to sign the consent form.
* Have already been included in the study previously.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 204 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Duration of crying in seconds | Through study completion, an average 6 months
  The duration of crying will be used as surrogate endpoint to assess pain

SECONDARY OUTCOMES:
The satisfaction of parents | Through study completion, an average 6 months
  The satisfaction of parents will be evaluated through a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil